CLINICAL TRIAL: NCT06744452
Title: App-based Stress Management: a Pragmatic Randomized Controlled Trial on the Efficacy of the MHealth Application "harmony"
Brief Title: App-based Stress Management with the MHealth Application "harmony"
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Witten/Herdecke (Other)
Responsible Party: Principal Investigator, Christina Hunger-Schoppe, Prof. Dr., University of Witten/Herdecke
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HARMONY RCT
Record Dates: First submitted 2024-09-09; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Stress; Self Efficacy; Resilience, Psychological; Goal Achievement; Well-Being, Psychological
Keywords: Stress management; Stress prevention; Application; App-based prevention
MeSH Terms: conditions — Psychological Well-Being | interventions — Harmony Hard

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- App-usage across a 12 week time period (Experimental): Use of the harmony application, with 6- and 12-week follow-up. Measurements will be taken at baseline as well as at 6- and 12-week follow-up.
  Interventions: Behavioral: harmony
- Waitlist-control group (No Intervention): Use of the harmony application after a 12-week waiting period. Measurements will be taken at baseline as well as at 6- and 12-week follow-up.

INTERVENTIONS:
Behavioral: harmony — Use of the app-based digital self-help intervention harmony over a 12-week-period. The app was designed for stress management and the preventive promotion of mental health. Harmony provides users with access to a wide range of psychological self-help content, including video episodes, audio sessions, texts, and downloadable materials. Utilizing artificial intelligence, Harmony offers personalized content suggestions tailored to the user's individual situation and preferences, ensuring the content remains relevant and updated. Content is delivered through a combination of psychoeducation, guided exercises, relaxation techniques, meditations, practical tasks, self-reflection activities, and everyday application tasks.
  Arms: App-usage across a 12 week time period

SUMMARY:
The purpose of this study is to investigate the efficacy of app-based stress prevention via the harmony application in a prospective, interventive, monocentric, explanatory pilot randomized controlled trial (RCT), with participants' subjective stress experience as the primary endpoint.

Research question: Does usage of the app harmony have a positive impact on the subjective experience of stress of its users? Do usage frequency, intensity or width of content engagement influence the efficacy of the intervention?

Hypothesis: We expect improvement of participants' subjective stress experience, stress-related symptoms, subjective well-being, resilient coping, self-efficacy, life satisfaction and goal-attainment.

ELIGIBILITY:
Inclusion Criteria:

* Increased stress level (PSS-10 >= 19; corresponds to one standard deviation (SD 6.42)) above the mean (PSS-10 = 12.57) in a representative sample of the German population (Klein et al., 2016)
* Fulfillment of technical minimum requirements (internet and smartphone access with suitable operating systems)
* German language skills at a native level or the ability to use the language at at least B level
* Written informed consent to participate in the study after being informed about the study

Exclusion Criteria:

* Inclusion criteria not met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2024-12-16 (Estimated); Primary Completion 2025-02-21 (Estimated); Study Completion 2025-02-21 (Estimated)

PRIMARY OUTCOMES:
Change from baseline stress at 6 weeks and 12 months | Baseline, 6-week follow-up, 12-week follow-up
  Perceived Stress Scale (PSS-10, Cohen et al., 1983): Self-report measure to assess psychological stress levels; Likert scale: 1 = never, 5 = very often.
Change from baseline stress symptoms at 6 weeks and 12 months | Baseline, 6-week follow-up, 12-week follow-up
  Stress and Coping Inventory (SCI; Satow, 2024): Self-report measure to assess psychological and physical stress symptoms; Likert scale: 1 = completely true (negative), 4 = not true at all (positive)

SECONDARY OUTCOMES:
Subjective well-being | Baseline, 6-week follow-up, 12-week follow-up
  WHO-5 Well-Being Index (WHO-5; WHO, 1998): Self-report measure to assess subjective well-being. Likert scale from 0 = at no time to 5 = all of the time.
Resilient coping | Baseline, 6-week follow-up, 12-week follow-up
  Brief resilient coping scale (BRCS; Kocalevent et al., 2014): Self-report measure to assess an individual's ability to cope with stress in a resilient manner. Likert scale from 1 = describes me not at all to 5 = describes me very well.
Self-efficacy | Baseline, 6-week follow-up, 12-week follow-up
  General Self-Efficacy Scale (GSE-SI; Di et al., 2023): One-item self-report measure to assess an individual's belief in their ability to perform tasks and handle situations effectively across a variety of contexts.
Life satisfaction | Baseline, 6-week follow-up, 12-week follow-up
  Life Satisfaction Scale (L-1; Beierlein et al., 2015): One-item self-report measure to assess a person's subjective evaluation of their quality of life. Likert scale from 1 = not satisfied at all to 11 = completely satisfied.
Goal Attainment | Baseline, 6-week follow-up, 12-week follow-up
  Goal Attainment Scaling (GAS; Grosse Holtforth & Grawe, 2002): Self-report measure to assess participants' previously set goals and their achievement; Scale from 0% to 100% in steps of 10%
Experience in Social Systems (EXIS; Hunger et al., 2017) | Baseline, 6-week follow-up, 12-week follow-up
  Self-report measure to assess systemic functioning in private and organizational social systems; Likert scale: 1 = not at all (negative), 6 = fully (positive)

OTHER OUTCOMES:
Frequency of application use | 6-week follow-up, 12-week follow-up (experiment group only)
  Participants' self report on absolut app usage over the past 6 weeks in days.
Duration of application use | 6-week follow-up, 12-week follow-up (experiment group only)
  Participants' self report on average app usage in minutes per session.
Extent of application use | 6-week follow-up, 12-week follow-up (experiment group only)
  Participants' self report on the extent of usage of different features within the app over the past six weeks. Respondents are asked to indicate which of the following functions they have used: Video, meditation, resilience course, texts, downloadable materials, and mental health checkup. Additionally, respondents specify the frequency of usage for each function.
User experience | 6-week follow-up, 12-week follow-up (experiment group only)
  Participants' self-report on overall impressions of the app. Likert scale from 1 = don't agree at all to 5 = completely agree
User satisfaction | 6-week follow-up, 12-week follow-up (experiment group only)
  Participants' self report on overall satisfaction with their experience using the app. Likert scale from 1 = very bad to 5 = very good

CONTACTS AND LOCATIONS:
Overall Officials: Christina Hunger-Schoppe, Prof. Dr., Study Director — University of Witten/Herdecke
Locations (1):
- Witten/Herdecke University, Witten, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Apolinario-Hagen J, Hennemann S, Fritsche L, Druge M, Breil B. Determinant Factors of Public Acceptance of Stress Management Apps: Survey Study. JMIR Ment Health. 2019 Nov 7;6(11):e15373. doi: 10.2196/15373. PMID 31697243